CLINICAL TRIAL: NCT07340320
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Dose-Finding Study of CX11 Tablets in Patients With Type 2 Diabetes Mellitus
Brief Title: A Study of CX11 Tablets in Patients With Type 2 Diabetes Mellitus
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Corxel Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CX11202
Record Dates: First submitted 2026-01-13; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Type II Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus; HbA1C; Percentage change in HbA1C; Change in Fasting Plasma Glucose; Change in body weight; Body weight loss; Hypoglycemics episodes; Hypoglycemia; Continuous Glucose Monitoring; Blood glucose; Health Survey Short Form-36; Diabetes treatment satisfaction questionnaire; Columbia-suicide severity rating scale
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypoglycemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Placebo group (Placebo Comparator)
  Interventions: Other: Placebo
- 40 mg group (Experimental)
  Interventions: Drug: CX11
- 80 mg group (Experimental)
  Interventions: Drug: CX11
- 120 mg group (Experimental)
  Interventions: Drug: CX11
- 160 mg group (Experimental)
  Interventions: Drug: CX11
- 200 mg group (Experimental)
  Interventions: Drug: CX11

INTERVENTIONS:
Drug: CX11 — CX11 tablets administered orally once daily (QD)
  Other Names: VCT220
  Arms: 120 mg group; 160 mg group; 200 mg group; 40 mg group; 80 mg group
Other: Placebo — Matching placebo tablets administered orally once daily (QD)
  Arms: Placebo group

SUMMARY:
This study is testing whether a new medication called CX11 works and is safe for participants with type 2 diabetes who have not reached good blood sugar control while taking a steady dose of metformin, with or without a steady dose of an SGLT2 inhibitor, for at least 90 days.

The study is being done at multiple medical centers. Participants are assigned by chance (randomized) to different groups, and neither the participants nor the study staff know which group they're in (double-blind). The groups are compared side by side (parallel), and some participants will receive inactive pills (placebo) to help measure the true effect of the study drug.

After screening, participants will be randomly placed into one of six groups, with equal chances of being in any group. Each group will receive a different dose of CX11 or a placebo. Treatment will last 24 weeks. After that, all participants will have a 2-week follow-up period to check on safety.

ELIGIBILITY:
Inclusion Criteria

Participants who meet all of the following criteria will be eligible to participate in this study:

* Adults aged 18 to 75.
* Diagnosis of type 2 diabetes for at least 6 months.
* HbA1c between 7.0% and 10.5%.
* Body mass index (BMI) between 23 and 50 kg/m².
* Body weight stable for the past 3 months before joining.
* Stable dose of metformin, with or without a stable dose of an SGLT2 inhibitor, for at least 3 months.
* Individuals who could become pregnant or could father a child must be willing and able to use highly effective birth control.

Exclusion Criteria

Participants who meet any of the following criteria will be excluded from this study:

* Type 1 diabetes or a history of diabetic ketoacidosis.
* Use of any GLP-1 receptor agonist within the past 6 months, or any prior exposure to CX11.
* Use of insulin to control blood sugar within the past 12 months.
* More than one episode of severe low blood sugar, with awareness of hypoglycemia symptoms.
* Cardiovascular or cerebrovascular conditions within the past 6 months:

  * Heart attack, coronary angioplasty, or bypass surgery (diagnostic angiography allowed).
  * Valvular heart disease or prior heart valve repair surgery.
  * Unstable angina.
  * Transient ischemic attack (TIA) or stroke.
  * Decompensated heart failure (NYHA Class III or IV).
  * ECG abnormalities indicating significant safety risk, such as supraventricular tachycardia, torsades de pointes, second- or third-degree AV block, myocardial infarction, QTcF > 450 ms in males or > 470 ms in females, PR interval > 220 ms.
  * Poorly controlled hypertension at screening: systolic ≥ 180 mmHg or diastolic ≥ 100 mmHg.
* Pancreatic or gallbladder conditions:

  * Acute or chronic pancreatitis.
  * Symptomatic gallbladder disease.
  * Pancreatic injury or risk factors that increase pancreatitis risk.
* Thyroid conditions:

  * Poorly controlled abnormal thyroid function on a stable dose before screening.
  * Clinically significant abnormal thyroid test results at screening.
  * Personal or first-degree family history of medullary thyroid carcinoma or multiple endocrine neoplasia (MEN) type 2A or 2B.
* Cancer history:

  * Malignancy within the past 5 years, regardless of recurrence or metastasis. Exceptions: localized basal cell skin cancer, low-risk prostate cancer, cervical carcinoma in situ, or high-grade prostatic intraepithelial neoplasia.
* Gastrointestinal conditions or treatments that may affect drug absorption:

  * Abnormal gastric emptying (e.g., gastric outlet obstruction).
  * Severe chronic gastrointestinal disease, including active ulcer within 6 months.
  * Crohn's disease, ulcerative colitis, or other inflammatory bowel diseases.
  * Prior gastrointestinal surgery (except polypectomy and appendectomy).
  * Long-term use of drugs that directly affect gastrointestinal motility (e.g., mosapride, cisapride).
* Liver disease:

  * Active liver disease other than nonalcoholic fatty liver.
  * Chronic active hepatitis B or C.
  * Primary biliary cirrhosis.
* Eye disease:

  * Uncontrolled or potentially unstable diabetic retinopathy or maculopathy.
* Abnormal lab results at screening:

  * eGFR < 60 mL/min/1.73 m² (CKD-EPI).
  * ALT or AST > 2.5 × upper limit of normal (ULN).
  * Total bilirubin > 1.5 × ULN (except known Gilbert's syndrome).
  * Serum amylase or lipase > 1.5 × ULN.
  * Fasting triglycerides > 5.7 mmol/L.
  * TSH > 1.5 × ULN.
  * Calcitonin ≥ 20 ng/L.
  * Hemoglobin < 110 g/L (male) or < 100 g/L (female).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2026-02-05 (Estimated); Primary Completion 2026-12-23 (Estimated); Study Completion 2027-01-07 (Estimated)

PRIMARY OUTCOMES:
Change in Glycosylated hemoglobin, Type A1C (HbA1c) from baseline | At Week 24

SECONDARY OUTCOMES:
Proportion of participants achieving HbA1c < 7.0% | At Week 24
Proportion of participants achieving HbA1c ≤ 6.5% | At Week 24
Change from baseline in Time in Range (TIR) measured by Continuous Glucose Monitoring (CGM) | To Week 24
Change from baseline in fasting plasma glucose (FPG) | To Week 24
Change in body weight from baseline | To Week 24
Percent change in body weight from baseline | To Week 24
Proportion of participants achieving body weight loss ≥ 5% | At Week 24
Proportion of participants achieving body weight loss ≥ 10% | At Week 24
Change in Systolic Blood Pressure (SBP) from baseline | To Week 24
Change in Diastolic Blood Pressure (DBP) from baseline | To Week 24
Number of Level 2 hypoglycemic episodes (glucose <54 mg/dL) | To Week 24
Number of severe hypoglycemic episodes | To Week 24
Number of treatment-emergent adverse events (TEAEs) | Study duration, approximately 26 weeks
Number of AEs of special interest (AESIs) | Study duration, approximately 26 weeks
Plasma drug concentrations at each specified sampling time point | At Weeks 2, 4, 6, 8, 12, 16, 22 and 24
Mean plasma drug concentration at each specified sampling time point | At Weeks 2, 4, 6, 8, 12, 16, 22 and 24

CONTACTS AND LOCATIONS:
Locations (46):
- United States (30):
  - Central Research Associates - Flourish - PPDS, Birmingham, Alabama
  - AES - DRS - Synexus Clinical Research US, Inc. - Birmingham, Birmingham, Alabama
  - AES - DRS - Optimal Research Alabama - Huntsville, Huntsville, Alabama
  - Ark Clinical Research - Long Beach, Long Beach, California
  - Flourish Research - Walnut Creek - PPDS, Walnut Creek, California
  - AES - DRS - Optimal Research Florida - Melbourne, Melbourne, Florida
  - Tampa General Hospital, Tampa, Florida
  - Conquest Research LLC - Winter Park, Winter Park, Florida
  - Privia Medical Group Georgia, LLC - Albany - Javara - PPDS, Albany, Georgia
  - Privia Medical Group Georgia, LLC - Savannah - Javara - PPDS, Savannah, Georgia
  - Privia Medical Group Georgia, LLC - Thomasville - Javara - PPDS, Thomasville, Georgia
  - AES - DRS - Synexus Clinical Research US, Inc. - Chicago, Chicago, Illinois
  - AES - DRS - Synexus Clinical Research US, Inc. - Evansville, Evansville, Indiana
  - Privia Medical Group, LLC - Kelly's Collaborative Care - Javara - PPDS, Silver Spring, Maryland
  - Elixia Health - Springfield - Elixia - PPDS, Springfield, Massachusetts
  - Elixia Health - Michigan Kidney Consultants, LLC - Elixia - PPDS, Pontiac, Michigan
  - AES - DRS - Synexus Clinical Research US, Inc. - Edina - Minneapolis, Edina, Minnesota
  - Mankato Clinic - East Main Street - Javara - PPDS, Mankato, Minnesota
  - Hassman Research Institute - Berlin - CenExel - PPDS, Berlin, New Jersey
  - Albuquerque Clinical Trials Inc, Albuquerque, New Mexico
  - M3 Wake Research, Inc - M3 WR, Raleigh, North Carolina
  - Unity Clinical Research, Oklahoma City, Oklahoma
  - Monroe Biomedical Research Charleston, North Charleston, South Carolina
  - M3 Wake Research - Dallas, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - SMS Clinical Research, LLC - 400 W. Kearney St, Mesquite, Texas
  - AES - DRS - Synexus Clinical Research US, Inc. - San Antonio, San Antonio, Texas
  - Flourish Research - San Antonio - PPDS, San Antonio, Texas
  - Privia Medical Group- North Texas - Stephenville - Javara - PPDS, Stephenville, Texas
  - Conquest Research - Arlington, Arlington, Virginia
- Poland (16):
  - AES - DRS - Synexus Polska Sp. z o.o. Oddzial w Poznaniu, Poznan, Greater Poland Voivodeship
  - Centrum Medyczne Pratia Bydgoszcz - PPDS, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Medyczne Centrum Diabetologiczno-Endokrynologiczno-Metaboliczne, Krakow, Lesser Poland Voivodeship
  - FutureMeds - Krakow - PPDS, Krakow, Lesser Poland Voivodeship
  - Gabinet Lekarski Robert Witek, Tarnów, Lesser Poland Voivodeship
  - METABOLICA Sp. z o.o, Tarnów, Lesser Poland Voivodeship
  - AES - DRS - Synexus Polska Sp. z o.o. Oddzial we Wroclawiu, Wroclaw, Lower Silesian Voivodeship
  - AES - DRS - Synexus Polska Sp. Z o.o. Oddzial w Lodzi, Lodz, Lódzkie
  - FutureMeds - Lodz - PPDS, Lodz, Lódzkie
  - FutureMeds - Warszawa Centrum - PPDS, Warsaw, Masovian Voivodeship
  - AES - DRS - Synexus Polska Sp. z o.o. Oddzial w Warszawie, Warsaw, Masovian Voivodeship
  - ETG Warszawa - PPDS, Warsaw, Masovian Voivodeship
  - AES - DRS - Synexus Polska Sp. z o.o. Oddzial w Gdansku, Gdansk, Pomeranian Voivodeship
  - AES - DRS - Synexus Polska Sp. z o.o. Oddzial w Gdyni, Gdynia, Pomeranian Voivodeship
  - AES - DRS - Synexus Polska Sp. z o.o. Oddzial w Czestochowie, Częstochowa, Silesian Voivodeship
  - AES - DRS - Synexus Polska Sp. z o.o. Oddzial w Katowicach, Katowice, Silesian Voivodeship

IPD SHARING:
Plan to Share IPD: No